CLINICAL TRIAL: NCT06908239
Title: Milk Temperature Control and Necrotizing Enterocolitis Risk in Extremely Preterm Infants: a Randomized Trial
Brief Title: Milk Temperature Control and Necrotizing Enterocolitis Risk in Extremely Preterm Infants
Acronym: NEC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other); children and women' hospital of Jiangxi (Unknown); Women and Children's Health Hospital of Qujing (Other); Guiyang Maternal and Child Health Care Hospital (Other); Maternal and Child Health Hospital of Guangxi Zhuang Autonomous Region (Other); Chengdu Women's and Children's Central Hospital (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Liuzhou Maternity and Child Healthcare Hospital (Other); Chongqing Medical Center for Women and Children (Other); Hunan children and women' hospital (Unknown)
Responsible Party: Principal Investigator, Chen Long,MD, director, Chongqing Medical Center for Women and Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Milk Temperature and NEC; 2024049 (Registry Identifier: Milk Temperature and NEC)
Record Dates: First submitted 2025-03-20; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-09

CONDITIONS: Necrotizing Enterocolitis; Preterm
Keywords: Necrotizing enterocolitis; preterm
MeSH Terms: conditions — Enterocolitis, Necrotizing; Premature Birth

STUDY DESIGN:
Intervention Model Description: In the thermostatic feeding group (intervention arm), milk or formula was delivered directly into the stomach via an infusion pump (Model 8713030CN, Shenzhen Shengnuo Medical Equipment Co., Ltd., Shenzhen, Guangdong, China) located within the incubator. The initial temperature of the milk was set at 38°C, and naturally decreased to match that of the incubator, maintaining a stable, thermostatic environment until the completion of feeding, as well as the setting and adjustment of the temperature of incubator according to the Chinese Medical Association guidelines
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- thermostatic feeding (Experimental): In the thermostatic feeding group (intervention arm), milk or formula was delivered directly into the stomach via an infusion pump (Model 8713030CN, Shenzhen Shengnuo Medical Equipment Co., Ltd., Shenzhen, Guangdong, China) located within the incubator. The initial temperature of the milk was set at 38°C, and naturally decreased to match that of the incubator, maintaining a stable, thermostatic environment until the completion of feeding, as well as the setting and adjustment of the temperature of incubator according to the Chinese Medical Association guidelines
  Interventions: Other: thermostatic feeding
- control (Active Comparator): In the control arm, standard feeding involved delivering breast milk or formula directly into the stomach using an infusion pump (Model 8713030CN) placed on an infusion stand. The initial temperature of the milk or formula was set at 38°C, and the temperature was allowed to naturally decrease to match the ambient air temperature of the NICU until feeding was completed. For both groups, the feeding volume and speed were managed in accordance with the clinical application guidelines for neonatal nutrition support in China.
  Interventions: Other: control

INTERVENTIONS:
Other: thermostatic feeding — In the thermostatic feeding group (intervention arm), milk or formula was delivered directly into the stomach via an infusion pump (Model 8713030CN, Shenzhen Shengnuo Medical Equipment Co., Ltd., Shenzhen, Guangdong, China) located within the incubator. The initial temperature of the milk was set at 38°C, and naturally decreased to match that of the incubator, maintaining a stable, thermostatic environment until the completion of feeding, as well as the setting and adjustment of the temperature of incubator according to the Chinese Medical Association guidelines
  Arms: thermostatic feeding
Other: control — In the control arm, standard feeding involved delivering breast milk or formula directly into the stomach using an infusion pump (Model 8713030CN) placed on an infusion stand. The initial temperature of the milk or formula was set at 38°C, and the temperature was allowed to naturally decrease to match the ambient air temperature of the NICU until feeding was completed. For both groups, the feeding volume and speed were managed in accordance with the clinical application guidelines for neonatal nutrition support in China.
  Arms: control

SUMMARY:
Necrotizing enterocolitis (NEC) is one of the most common and severe gastrointestinal emergencies during the neonatal period, especially among preterm infants. In high-income countries such as Finland and the USA, the prevalence of NEC ranges from 2% to 16.58% among very preterm infants (VPIs) and from 6.8% to 10.0% among extremely preterm infants (EPIs). According to the 2022 Annual Report of the China Newborn Collaboration Network (CHNN) from 89 tertiary hospitals, the prevalence of NEC was reported at 14.2% among VPIs and EPIs. Up to half of NEC cases in infants require surgical intervention, with 39.1% of VPIs and 44.5% of EPIs needing surgery. Consequently, NEC-related mortality rates vary significantly, ranging from 21.9% to 42.3% in preterm infants weighing less than 1500 grams (equivalent to VPIs) and from 33.0% to 50.5% in those weighing 500-1000 grams (equivalent to EPIs).

DETAILED DESCRIPTION:
Although the pathophysiology of NEC is not fully understood, epidemiological studies strongly suggest a multifactorial cause, involving infection and inflammation, premature birth, hypoxic-ischemia, improper feeding, and cold exposure. As for cold exposure, it encompasses inhaling cold air through the respiratory tract, contact with cold environments through the skin, and consuming cold food through the digestive tract. Such exposure increases the risks of cardiovascular hospitalization, temperature-related mortality, allergic diseases including asthma and atopic dermatitis, and neonatal death. A recent study by Lyu et al. suggested that admission hypothermia is associated with an increased incidence of NEC. However, no research has systematically explored how preventing cold exposure, such as through milk feeding via the digestive tract, could potentially reduce the development of NEC among EPIs/VPIs.

Covariates collected using medical records throughout study conduction included maternal age, neonatal sex, birthweight and gestational age at delivery, and weekly weight until discharged. Gestational diabetes mellitus was diagnosed based on a 2-hour 75g three-time-point oral glucose tolerance test was performed at the clinic according to the International Association of Diabetes and Pregnancy Study (IADPSG) criteria adopted by Chinese Obstetrics and Gynecology guidelines between 24 and 28 weeks of gestation. The investigators collected information on clinical diagnosis of hypertension disorders during pregnancy (HDP) from medical records, which was defined by systolic blood pressure (SBP) ≥140 mm Hg and/or diastolic blood pressure (DBP) ≥ 90 mm Hg, with positive proteinuria, at any timepoints between week 20 and delivery.Other pregnancy outcomes or complications were also retrieved from the medical databased, such as the admission of antenatal corticoids, placenta previa, premature rupture of the membrane, and intrahepatic cholestasis of pregnancy that were diagnosed based on national guidelines. As for infants, neonatal critical case score (NCIS) were assessed within 24 hours of admission and divided into non-critical group (>90), critical group (70-90) and extremely critical group (<70) according to the Chinese Pediatric guidelines. Others neonatal medical conditions during hospitalization were also recorded if diagnosed based on international guidelines, namely small-for-gestational age (SGA), respiratory distress syndrome (RDS) and early onset of sepsis (EOS) within three days after birth. In addition, the days to diagnosis of NEC, length of stay during hospitalization, and cases of surgery among NEC cases were collected from thermostatic feeding and standard feeding groups.

ELIGIBILITY:
Inclusion Criteria:

* gestational age at delivery between 24+0 and 31+6 weeks
* initiation of enteral nutrition within 24 hours after birth.

Exclusion Criteria:

* parental decision to not participate
* presence of major congenital anomalies
* requirement for surgical intervention prior to randomization.

The subject would be considered censored if the study ended due to one of the following conditions:

* 1. Death
* 2. Parents' decision to withdraw participation
* 3. Discharge based on doctors' recommendations.

Once enrolled, the neonates received minimal enteral nutrition within the first 24 hours after birth for the initial three days. Following this period, both groups of neonates were fed expressed milk using a pumping system.

the milk temperature was measured using the following steps:

* 1) During the first week after birth, each preterm infant had two identical pumping setups. One pump was used for feeding according to group allocation, while the second, set to zero velocity, was used to measure milk temperature
* 2) The temperature from the second pump, taken at the same time milk entered the stomach from the first pump, was recorded as the final milk temperature
* 3) After the first week, only one pump was used per infant, and the temperature of the last 1 ml of milk was measured as the final temperature.

Both groups were supplemented with human milk fortifier (HMF) for preterm infants weighing 1800 g or less. The neonates were fed 50 ml/kg/day of breast milk, following the Chinese Expert Consensus on the Use of Breast Milk Fortifiers in Premature Infants. The milk was sourced from the infant's mother. Initially, infants received half-strength fortified milk for 3-7 days before transitioning to full-strength fortified milk. HMF was discontinued once the infant's body weight reached the 25th-50th percentile for appropriate-for-gestational-age infants or the 10th percentile for small-for-gestational-age infants, depending on sex and gestational age. The choice of formula, HMF, and the decision to add lactase was at the discretion of the attending neonatologist.

Weaning from thermostatic feeding would occur if any of the following conditions were met:

* 1) If no signs of feeding intolerance (FI) appeared after administering pumped milk within 15 minutes for 1-2 days, thermostatic feeding would transition to standard feeding
* 2) The feeding duration could be gradually reduced in 10-minute increments down to a minimum of 15 minutes. Weaning from standard feeding would occur if no FI was observed after oral feeding within 30 minutes for 1-2 days.

Due to the lack of existing intervention-based evidence for reference, we based our sample size calculation on an RCT that examined the impact of feeding patterns (human milk-based diet vs. bovine milk-based products). According to the published data, the incidence of NEC was significantly lower in infants receiving an exclusively human-milk-based diet (4.5%) compared to those receiving bovine milk-based products (15.9%; p = 0.04), with approximately 10% in difference of incidence. Using previously published data on NEC prevention, we conducted a power analysis for a superiority clinical trial. To achieve 80% power with a 5% Type I error rate (α = 0.05), we estimated a sample size of 100 participants per group (n₁ = 100, n₂ = 100). Considering a 20% loss to follow-up, we adjusted the sample size to 120 participants per group to ensure adequate power to detect an approximately 10% difference in NEC incidence between the intervention and control groups (R version 4.2.2).

Ages: 24 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of necrotizing enterocolitis (NEC) | three months after admission
  Primary outcome was the incidence of necrotizing enterocolitis (NEC), specifically focusing on cases classified as Bell's stage ≥2, according to the modified Bell's staging criteria for NEC

SECONDARY OUTCOMES:
the incidence of bronchopulmonary dysplasia(BPD) | at 36 weeks' gestational age
  Bronchopulmonary dysplasia (BPD) was diagnosed at a corrected gestational age of 36 weeks, following the NICHD definition established in 2019
the incidence of late-on sepsis(LOS) | three months after admission
  Late-onset sepsis (LOS) was defined by the expert consensus on the diagnosis and management of neonatal sepsis (version 2019) with onset beyond three days after admission
the incidence of intraventricular hemorrhage(IVH) | three months after admission
  Intraventricular hemorrhage (IVH) was presented with grades 1-4.
the incidence of retinopathy of Prematurity(ROP) | three months after admission
  Retinopathy of prematurity (ROP) was categorized according to the International Classification of Retinopathy of Prematurity, revised in 2005
the incidence of hematochezia | three months after admission
  Hematochezia was presented and diagnosed
the incidence of extra-uterine growth restriction(EUGR) | at 36 weeks' corrected gestational age
  Extrauterine growth retardation (EUGR) was identified at a corrected gestational age of 36 weeks, based on the Fenton growth chart for preterm infants

CONTACTS AND LOCATIONS:
Overall Officials: Long Long, MD.,PhD, Principal Investigator — Women and Children's Hospital of Chongqing Medical University
Locations (1):
- Chongqing Health Center for Women and Children, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
patients data after paper published after request
Supporting Information: Study Protocol, SAP
Time Frame: patients data after paper published after request for three months
Access Criteria: Doctor Long Chen. patients' data after request